CLINICAL TRIAL: NCT01715818
Title: A PHASE 3B STUDY TO EVALUATE THE POTENTIAL OF ALEGLITAZAR TO REDUCE CARDIOVASCULAR RISK IN PATIENTS WITH STABLE CARDIOVASCULAR DISEASE AND GLUCOSE ABNORMALITIES
Brief Title: A Study on The Potential of Aleglitazar to Reduce Cardiovascular Risk in Patients With Stable Cardiovascular Disease and Glucose Abnormalities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC28027; 2012-000671-16 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Disease, Diabetes Mellitus Type 2
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — matching aleglitazar placebo tablet orally daily
  Arms: Placebo
Drug: aleglitazar — 150 mcg orally daily
  Arms: Aleglitazar

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group, multicenter study will evaluate the potential of aleglitazar to reduce cardiovascular risk in patients with stable cardiovascular disease and glucose abnormalities. Patients will be randomized 1:1 to receive either aleglitazar 150 mcg orally daily or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with established evidence of stable cardiovascular disease (CVD) defined as at least one of the following groups of criteria (A or B) A. Age >/= 40 years with history with prior CV event of prior myocardial infarction or prior ischemic stroke (confirmed by brain imaging study), with onset >/= 3 months prior to randomization and stable in the Investigator's judgment B. Age >/= 55 years with evidence of CVD (stable in the Investigator's judgment), defined as at least one of the following: Coronary disease, cerebrovascular disease or peripheral arterial disease as defined by protocol
* Patients with glucose abnormalities based on one of the following A-B criteria:

A. Established Type 2 diabetes mellitus (T2D) according to 2010 ADA criteria; treatment may include diet alone, or any glucose-lowering therapies except for thiazolidinediones (TDZs) B. No fulfillment of criterion A) but evidence of glucose abnormalities

* Optimal management of CV risk factors including hypertension and dyslipidemia as informed by the best evidence and clinical practice guidelines

Exclusion Criteria:

* Current treatment with a thiazolidinedione (TDZ) or fibrate
* Prior intolerance to a TDZ or fibrate
* Previous participation in a trial with aleglitazar
* Other types of diabetes
* Inadequate liver, hematologic or renal function
* Symptomatic heart failure classified as NYHA class II-IV
* Hospitalization for a primary diagnosis of heart failure in the 12-month period preceding randomization
* Peripheral edema which in the judgment of the Investigator in believed to be severe and of cardiac origin
* History of surgical coronary revascularization (CABG) less than 5 years prior to screening, except in cases of subsequent myocardial infarction
* Currently scheduled for arterial revascularization procedures
* Systemic corticosteroid therapy for > 2 weeks within 3 months prior to screening
* Diagnosed or treated malignancy (except for treated basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) within the past 5 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1999 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of any component of the composite event (cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke) as adjudicated by the Clinical Events Committee (CEC) | 5 years

SECONDARY OUTCOMES:
Time to first occurrence of a composite with components as adjudicated by the CEC: cardiovascular death, non-fatal MI and non-fatal stroke (in each of the subgroups with or without evidence of T2D at baseline) | 5 years
Time to first occurrence of a composite with components as adjudicated by the CEC: all-cause mortality, non-fatal MI and non-fatal stroke (in each of the subgroups with or without evidence of T2D at baseline) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (312):
- United States (129):
  - Muscle Shoals, Alabama
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Cudahy, California
  - Encino, California
  - Fresno, California
  - Hawaiian Gardens, California
  - Huntington Beach, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - North Hollywood, California
  - Northridge, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - Stockton, California
  - Thousand Oaks, California
  - Torrance, California
  - Tustin, California
  - Ventura, California
  - Denver, Colorado
  - Atlantis, Florida
  - Bradenton, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Pinellas Park, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Dunwoody, Georgia
  - Eagle, Idaho
  - Idaho Falls, Idaho
  - Melrose Park, Illinois
  - Brownsburg, Indiana
  - Evansville, Indiana
  - Valparaiso, Indiana
  - Council Bluffs, Iowa
  - Iowa City, Iowa
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Alexandria, Louisiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Haverhill, Massachusetts
  - Traverse City, Michigan
  - Fall Rivers, Mississippi
  - Kansas City, Missouri
  - Bellevue, Nebraska
  - Fremont, Nebraska
  - Las Vegas, Nevada
  - Elizabeth, New Jersey
  - Albany, New York
  - North Massapequa, New York
  - Smithtown, New York
  - Syracuse, New York
  - Westfield, New York
  - Elizabeth City, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Shelby, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Gallipolis, Ohio
  - Kettering, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Doylestown, Pennsylvania
  - Fleetwood, Pennsylvania
  - Harleysville, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Uniontown, Pennsylvania
  - Clinton, South Carolina
  - Greer, South Carolina
  - Murrells Inlet, South Carolina
  - Varnville, South Carolina
  - Dakota Dunes, South Dakota
  - Chattanooga, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Kingwood, Texas
  - McAllen, Texas
  - New Braunfels, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Bountiful, Utah
  - Draper, Utah
  - Murray, Utah
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
  - Suffolk, Virginia
  - Port Orchard, Washington
  - Spokane, Washington
  - Madison, Wisconsin
- Caba, Argentina
- Australia (13):
  - Camperdown, New South Wales
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Wollongong, New South Wales
  - South Brisbane, Queensland
  - Adelaide, South Australia
  - Woodville, South Australia
  - Launceston, Tasmania
  - Geelong, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Armadale, Western Australia
  - Perth, Western Australia
- Austria (4):
  - Braunau am Inn
  - Feldkirch
  - Graz
  - Vienna
- Canada (27):
  - Kelowna, British Columbia
  - Surrey, British Columbia
  - Winnipeg, Manitoba
  - Bathurst, New Brunswick
  - Cambridge, Ontario
  - Collingwood, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Quebec, Prince Edward Island
  - Chicoutimi, Quebec
  - Granby, Quebec
  - Lachine, Quebec
  - Laval, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec
  - Terrebonne, Quebec
  - Saskatoon, Saskatchewan
- Chile (3):
  - Las Condes
  - Santiago
  - Temuco
- Colombia (6):
  - Barranquila
  - Barranquilla
  - Bogotá
  - Cartagena
  - Floridablanca
  - Medellín
- Czechia (8):
  - Beroun
  - Brno
  - Jihlava
  - Liberec
  - Prague
  - Praha 4 - Krc
  - Slaný
  - Třebíč
- Estonia (3):
  - Narva
  - Tallinn
  - Tartu
- Germany (18):
  - Berlin
  - Bochum
  - Charlottenburg
  - Chemnitz
  - Cologne
  - Damme
  - Dresden
  - Frankfurt
  - Hanover
  - Homburg/Saar
  - Kassel
  - Köthen
  - Leipzig
  - Magdeburg
  - Mönchengladbach
  - Münster
  - Neunkirchen
  - Wangen
- Hungary (11):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Gyöngyös
  - Mosonmagyaróvár
  - Nyíregyháza
  - Pápa
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Zalaegerszeg
- Giv‘atayim, Israel
- Italy (10):
  - Naples, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Pavia, Lombardy
  - Catania, Sicily
  - Palermo, Sicily
  - Pesaro, The Marches
  - Massa, Tuscany
- Tochigi, Japan
- Latvia (2):
  - Liepāja
  - Riga
- Lithuania (2):
  - Kaunas
  - Vilnius
- Malaysia (6):
  - Johor Bahru
  - Kuala Lumpur
  - Kuala Selangor
  - Perak
  - Sabak Bernam
  - Sarawak
- Mexico (5):
  - Aguascalientes
  - México
  - Monclova
  - Monterrey
  - Xalapa
- Poland (11):
  - Bialystok
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Nowy Sącz
  - Opole
  - Rzeszów
  - Warsaw
  - Wroclaw
- Romania (6):
  - Baia Mare
  - Bucharest
  - Craiova
  - Oradea
  - Ploieşti
  - Târgu Mureş
- Russia (3):
  - Kemerovo
  - Saint Petersburg
  - Tomsk
- South Africa (2):
  - Pretoria
  - Pretoria West
- South Korea (8):
  - Busan
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Seoul
  - Suwon
  - Wŏnju
- Spain (17):
  - Albacete, Albacete
  - Sant Joan d'Alacant, Alicante
  - Almería, Almeria
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Girona, Girona
  - Granada, Granada
  - Huelva, Huelva
  - Santiago de Compostela, La Coruña
  - Lleida, Lerida
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
  - Tarragona, Tarragona
  - Alzira, Valencia
  - Valencia, Valencia
- Sweden (2):
  - Malmo
  - Stockholm
- Thailand (2):
  - Bangkok
  - Khon Kaen
- United Kingdom (11):
  - Birmingham
  - Cardiff
  - Chorley
  - Edinburgh
  - Glasgow
  - Inverness
  - Liverpool
  - Manchester
  - Mortimer
  - Reading
  - Soham, Ely